CLINICAL TRIAL: NCT05954312
Title: A Phase 1, Open-label, Multicenter, First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Anti-tumor Activity of VVD-130037, a Kelch-like ECH Associated Protein 1 (KEAP1) Activator, in Participants With Advanced Solid Tumors
Brief Title: A First-in-Human (FIH) Study to Evaluate the Safety and Tolerability of VVD-130037 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vividion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VVD-130037-001; 2023-506199-28-00 (EU CTIS Number)
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors
Keywords: VVD-130037; First-in-Human; KEAP1; NRF2; Cancer; small molecule; squamous cell histology; esophageal adenocarcinoma
MeSH Terms: conditions — Neoplasms; Adenocarcinoma Of Esophagus | interventions — Docetaxel; Paclitaxel; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1 (Dose Escalation): VVD-130037 Single Agent (Experimental): Participants will receive ascending doses of VVD-130037, orally, once or twice daily in 21-day treatment cycles during Part 1.
  Interventions: Drug: VVD-130037
- Part 1 (Dose Escalation): VVD-130037 and Docetaxel Combination Therapy (Experimental): Participants will receive ascending doses of VVD-130037, orally, once or twice daily along with docetaxel intravenous (IV) infusion administered once every 3 weeks in 21-day treatment cycles during Part 1.
  Interventions: Drug: VVD-130037; Drug: Docetaxel
- Part 1 (Dose Escalation): VVD-130037 and Paclitaxel Combination Therapy (Experimental): Participants will receive ascending doses of VVD-130037, orally, once or twice daily along with paclitaxel IV infusion administered on Days 1, 8, and 15 of each 28-day treatment cycle during Part 1.
  Interventions: Drug: VVD-130037; Drug: Paclitaxel
- Part 2 (Dose Expansion): VVD-130037 Single Agent (Experimental): Participants will receive VVD-130037 at the recommended dose for expansion (RDE), orally, once or twice daily in 21-day treatment cycles during Part 2.
  Interventions: Drug: VVD-130037
- Part 2 (Dose Expansion): VVD-130037 and Docetaxel Combination Therapy (Experimental): Participants will receive VVD-130037 at the RDE, orally, once or twice daily along with docetaxel IV infusion administered once every 3 weeks in 21-day treatment cycles during Part 2.
  Interventions: Drug: VVD-130037; Drug: Docetaxel
- Part 2 (Dose Expansion): VVD-130037 and Paclitaxel Combination Therapy (Experimental): Participants will receive VVD-130037 at the RDE, orally, once or twice daily along with paclitaxel IV infusion administered on Days 1, 8, and 15 of each 28-day treatment cycle during Part 2.
  Interventions: Drug: VVD-130037; Drug: Paclitaxel
- Experimental: Part 2 (Dose Expansion): VVD-130037 and Pembrolizumab Combination Therapy (Experimental): Participants will first be evaluated in a safety-run in cohort to determine the RDE(s). Participants will then receive VVD-130037 at the RDE, orally, once or twice daily along with pembrolizumab IV infusion administered once every 3 weeks in 21-day treatment cycles during Part 2.
  Interventions: Drug: VVD-130037; Drug: Pembrolizumab

INTERVENTIONS:
Drug: VVD-130037 — Oral tablets
Drug: Docetaxel — IV infusion
  Arms: Part 1 (Dose Escalation): VVD-130037 and Docetaxel Combination Therapy; Part 2 (Dose Expansion): VVD-130037 and Docetaxel Combination Therapy
Drug: Paclitaxel — IV infusion
  Arms: Part 1 (Dose Escalation): VVD-130037 and Paclitaxel Combination Therapy; Part 2 (Dose Expansion): VVD-130037 and Paclitaxel Combination Therapy
Drug: Pembrolizumab — IV infusion
  Arms: Experimental: Part 2 (Dose Expansion): VVD-130037 and Pembrolizumab Combination Therapy

SUMMARY:
A FIH dose escalation and dose expansion study to evaluate VVD-130037 in participants with advanced solid tumors as a single agent, and in combination with docetaxel, paclitaxel, or pembrolizumab.

ELIGIBILITY:
Key Inclusion Criteria for Parts 1 and 2:

* Histologically or cytologically confirmed metastatic or unresectable solid tumor.
* Measurable disease by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as assessed by the Investigator.
* Have progressed on or after all prior standard-of-care therapies for metastatic disease.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
* Adequate organ and marrow function as defined in the protocol.

Additional Key Inclusion Criteria for Part 2:

* Participants with squamous non-small cell lung cancer (sqNSCLC) with or without nuclear factor erythroid 2-related factor 2 (NRF2 [NFE2L2]) and/or cullin 3 (CUL3) mutations.
* Participants with advanced sqNSCLC must be refractory to or have progressed on or after a platinum-based doublet regimen and an immune checkpoint inhibitor.
* Participants with advanced head and neck squamous cell carcinoma (HNSCC) must have received prior treatment with platinum-based chemotherapy, an immune checkpoint inhibitor (for tumors with known programmed death-ligand 1 [PD-L1] expression, microsatellite instability-high, or mismatch repair deficiency, and an anti-epidermal growth factor receptor agent) (Combination Expansion Cohort).
* Participants with advanced esophageal squamous cell carcinoma (ESCC) must have received prior treatment with platinum-based chemotherapy, an immune checkpoint inhibitor (for tumors with known PD-L1 expression) (Combination Expansion Cohort).
* Participants with a known driver mutation, including activating epidermal growth factor receptor mutations or anaplastic lymphoma kinase rearrangements, should have progressed after appropriate targeted treatment.
* Participants with known human epidermal growth factor receptor 2 overexpression should have progressed after appropriate targeted treatment.

Key Exclusion Criteria for Parts 1 and 2:

* Participant is known to have a mutation that has no expectation of benefit from VVD-130037. Current such mutations include the following:

  1. KEAP1 nonsense mutation (any position)
  2. KEAP1 frameshift mutation (any position)
* Any unresolved toxicity Grade ≥2 per CTCAE version 5.0 from previous anticancer treatment.
* Current or prior treatment with anti-epileptic medications for the treatment or prophylaxis of seizures.
* History of seizure or condition that may predispose to seizure.
* History or presence of central nervous system (CNS) metastases or spinal cord compression.
* Uncontrolled arterial hypertension despite optimal medical management.
* Risk factors for abnormal heart rhythm/QT prolongation as defined in the protocol.
* History of the following cardiac diseases:

  i) congestive heart failure (New York Heart Association [NYHA] Class >II), ii) unstable angina, iii) new onset angina within past 6 months, iv) myocardial Infarction within the past 6 months, v) clinically significant arrhythmias within past 6 months.
* Any prior toxicity (Grade 3 or 4) related to immunotherapy leading to treatment discontinuation (Combination Expansion Cohort)
* Medical history of (noninfectious) pneumonitis/interstitial lung disease (ILD), drug induced ILD, radiation pneumonitis that required steroid treatment, or any evidence of clinically active pneumonitis/ILD (Combination Expansion Cohort)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2030-08-31 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
Part 1 (Dose Escalation): Incidence and Severity of Dose-limiting Toxicities (DLTs) During DLT Observation Period | Part 1: Single Agent and Docetaxel/Pembrolizumab Combination Therapy: From Day 1 to Day 21 of Cycle 1 [cycle length=21 days] and Part 1: Paclitaxel Combination Therapy: From Day 1 to Day 28 of Cycle 1 [cycle length=28 days]
  Incidence and severity of DLTs will be assessed per DLT criteria set forth in the protocol based on adverse events (AEs) evaluated per National Cancer Institute (NCI) - Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Part 2 (Dose Expansion): Number of Participants With AEs, Serious Adverse Events (SAEs), and Clinical Laboratory Abnormalities | Up to approximately 4 years

SECONDARY OUTCOMES:
Part 1 (Dose Escalation): Number of Participants With AEs, SAEs, and Clinical Laboratory Abnormalities | Up to approximately 4 years
Part 2 (Dose Expansion): Recommended Phase 2 Dose (RP2D) of VVD-130037 as a Single Agent and in Combination with Docetaxel, Paclitaxel, or Pembrolizumab | Up to approximately 4 years
  The RP2D will be based on safety, tolerability, pharmacokinetics and preliminary anti-tumor activity of VVD-130037 as single agent, and in combination with docetaxel, paclitaxel, or pembrolizumab during Part 2.
Part 2 (Dose Expansion): Overall Response Rate (ORR) | Up to approximately 4 years
  ORR is defined as the percentage of participants achieving a best overall response of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator assessment.
Part 2 (Dose Expansion): Duration of Response (DOR) | Up to approximately 4 years
  DOR is defined as the time from initial response of CR or PR to progressive disease or death, whichever comes first per RECIST version 1.1 by investigator assessment.
Part 2 (Dose Expansion): Progression-free Survival (PFS) | Up to approximately 4 years
  PFS is defined as the time from the date of randomization to the time of confirmed disease progression or death, whichever occurs first per RECIST version 1.1 by investigator assessment.
Part 2 (Dose Expansion): Disease Control Rate (DCR) | Up to approximately 4 years
  DCR is defined as the percentage of participants achieving CR or PR, or stable disease (SD) per RECIST version 1.1 by investigator assessment.
Parts 1 and 2 (Dose Escalation and Expansion): Area Under the Plasma Concentration-time Curve (AUC) of VVD-130037 | Parts 1 and 2: Predose and multiple timepoints post-dose from Cycle 1 Day 1 up to Cycle 5 Day 1 (cycle length=21 days for Single Agent and Docetaxel/Pembrolizumab Combination Therapy and cycle length=28 days for Paclitaxel Combination Therapy)
Parts 1 and 2 (Dose Escalation and Expansion): Maximum Observed Concentration (Cmax) of VVD-130037 | Parts 1 and 2: Predose and multiple timepoints post-dose from Cycle 1 Day 1 up to Cycle 5 Day 1 (cycle length=21 days for Single Agent and Docetaxel/Pembrolizumab Combination Therapy and cycle length=28 days for Paclitaxel Combination Therapy)
Parts 1 and 2 (Dose Escalation and Expansion): Apparent Terminal Half-life (T1/2) of VVD-130037 | Parts 1 and 2: Predose and multiple timepoints post-dose from Cycle 1 Day 1 up to Cycle 5 Day 1 (cycle length=21 days for Single Agent and Docetaxel/Pembrolizumab Combination Therapy and cycle length=28 days for Paclitaxel Combination Therapy)
Parts 1 and 2 (Dose Escalation and Expansion): QT/Corrected QT (QTc) Interval and Other Electrocardiogram (ECG) Parameters | Parts 1 and 2: Up to approximately 4 years
  Number of participants with changes in QT/QTc interval and other ECG parameters will be assessed.

CONTACTS AND LOCATIONS:
Locations (25):
- United States (8):
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MDACC, Houston, Texas
  - NEXT Dallas, Irving, Texas
  - NEXT Virginia, Fairfax, Virginia
- South Korea (8):
  - National Cancer Center, Goyang
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University; Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital; Yonsei University Health System, Seoul
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon
- Spain (9):
  - Hospital Vall d'Hebron, Barcelona
  - START Barcelona Hospital HM Nou Delfos, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - NEXT Madrid, Madrid
  - START Madrid CIOCC, Madrid
  - Start Madrid-FJD, Hospital Fundacion Jimenez Diaz, Madrid
  - Clinica Universitaria de Navarra, Pamplona
  - Hospital Clinico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roy N, Wyseure T, Lo IC, Lu J, Eissler CL, Bernard SM, Bok I, Snead AN, Parker A, Lo UG, Green JC, Inloes J, Jacinto SR, Kuenzi B, Pariollaud M, Negri K, Le K, Horning BD, Ibrahim N, Grabow S, Panda H, Bhatt DP, Wilkerson EM, Saeidi S, Zolkind P, Rush Z, Williams HN, Walton E, Pastuszka MK, Sigler JJ, Tran E, Hee K, McLaughlin J, Ambrus-Aikelin G, Pollock J, Abraham RT, Kinsella TM, Simon GM, Major MB, Weinstein DS, Patricelli MP. A covalent allosteric molecular glue suppresses NRF2-dependent cancer growth. Cancer Discov. 2025 Dec 19. doi: 10.1158/2159-8290.CD-25-1187. Online ahead of print. PMID 41417010